CLINICAL TRIAL: NCT06680440
Title: A Phase I Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ASC30 Tablets in Participants With Obesity
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of ASC30 Tablets and ASC30 Tablets A1 in Participants With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascletis Pharma (China) Co., Limited (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASC30-102
Record Dates: First submitted 2024-10-30; First posted 2024-11-08 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-09

CONDITIONS: Weight Management

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- SAD Cohort 1 (Experimental): SAD dose 1
  Interventions: Drug: ASC30; Other: Placebo
- SAD Cohort 2 (Experimental): SAD dose 2
  Interventions: Drug: ASC30; Other: Placebo
- SAD Cohort 3 (Experimental): SAD dose 3
  Interventions: Drug: ASC30; Other: Placebo
- SAD Cohort 4 (Experimental): SAD dose 4
  Interventions: Drug: ASC30; Other: Placebo
- SAD Cohort 5 (Experimental): SAD dose 5
  Interventions: Drug: ASC30; Other: Placebo
- MAD Cohort 1 (Experimental): MAD dose 1
  Interventions: Drug: ASC30; Other: Placebo
- MAD Cohort 2 (Experimental): MAD dose 2
  Interventions: Drug: ASC30; Other: Placebo
- MAD Cohort 3 (Experimental): MAD dose 3
  Interventions: Drug: ASC30; Other: Placebo

INTERVENTIONS:
Drug: ASC30 — Tablet, QD
Other: Placebo — Tablets, QD

SUMMARY:
This is a phase I, randomized, double-blind, placebo-controlled, single and multiple ascending dose study to evaluate the safety, tolerability, pharmacokinetics, efficacy, food effect of ASC30 Tablets or ASC30 Tablets A1 in participants with obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided informed consent before initiation of any study-specific procedures.
2. Male or female participants, non-smokers, between 18 and 65 years of age (both inclusive).
3. No clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and other screening procedures.

Exclusion Criteria:

1. Have evidence of any clinically significant active or chronic disease.
2. Have any prior diagnosis of diabetes mellitus (T1DM or T2DM), or rare forms of diabetes mellitus.
3. Have an autoimmune disease, is immunosuppressed or is in any way immunocompromised.
4. Have a history of acute or chronic pancreatitis.
5. Participants with a known clinically significant gastric emptying abnormality.
6. Have a history of an active or untreated malignancy or are in remission from a clinically significant malignancy.
7. Have a history of any other condition (such as known drug or alcohol abuse, diagnosed eating disorder, or other psychiatric disorder) that, in the opinion of the Investigator, may preclude the participant from following and completing the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs, SAEs (Safety and Tolerability) of ASC30 (SAD) | Up to Day 8
  A summary of AEs, SAEs and other non-serious adverse events
Incidence of AEs, SAEs (Safety and Tolerability) of ASC30 (MAD) | Up to Day 28
  A summary of AEs, SAEs and other non-serious adverse events

SECONDARY OUTCOMES:
Cmax of ASC30 (SAD) | Up to Day 8
  PK parameters of ASC30
Cmax of ASC30 (MAD) | Up to Day 28
  PK parameters of ASC30
Change From Baseline in Body Weight (MAD) | Up to Day 28
  Change From Baseline in Body Weight

CONTACTS AND LOCATIONS:
Locations (1):
- Ascletis clinical site, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No